CLINICAL TRIAL: NCT05974124
Title: Topical Ophthalmic Antiseptics and Reduction of Ocular Surface Bacterial Load Before Cataract Surgery: a Randomized Clinical Trial
Brief Title: Effectiveness of Ophthalmic Antiseptic Preparations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: European School of Advanced Studies in Ophthalmology (Other)
Responsible Party: Principal Investigator, Vito Romano, Professor, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OS1
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Antiseptics; Microbiota; Conjunctiva
Keywords: Povidone-iodine; Chlorhexidine; Preoperative; Antiseptics; Conjunctival bacterial flora

STUDY DESIGN:
Intervention Model Description: Participants were randomised to instill either povidone-iodine eye drops (35 patients) or chlorhexidine (35 patients) in the eye to be operated on. The contralateral eye was considered as control and received no antiseptic prophylaxis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Povidone-Iodine 0.66%
  Interventions: Device: Povidone-Iodine 0.66%
- Group B (Experimental): Chlorhexidine 0.02%
  Interventions: Device: Chlorhexidine 0.02%

INTERVENTIONS:
Device: Povidone-Iodine 0.66% — Povidone-iodine 0.66% eye drops were instilled 4 times daily for 3 days before cataract surgery in the eye to be operated on. The contralateral eye was considered as control and received no treatment.
  Arms: Group A
Device: Chlorhexidine 0.02% — Chlorhexidine 0.02% eye drops were instilled 4 times daily for 3 days before cataract surgery in the eye to be operated on. The contralateral eye was considered as control and received no treatment.
  Arms: Group B

SUMMARY:
The aim of this clinical trial is to evaluate the effectiveness of two topical antiseptics, povidone-iodine (PVI) and chlorhexidine (CHX), in reducing conjunctival bacterial flora.

DETAILED DESCRIPTION:
70 patients undergoing cataract surgery were enrolled and randomly divided in two arms: 35 patients used PVI 0.66% 4 times daily starting 3 days before surgery; 35 patients used CHX 0.02% with the same posology. The contralateral eye was considered as control. Conjunctival swabs were collected in both eyes at the baseline (T0) and after three days of treatment (T1) all before cataract surgery. Conjunctival bacterial load has been evaluated through a molecular based method at T0 and T1 and compared to the control eye.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cataract surgery
* 18 years of age or older

Exclusion Criteria:

* Reported allergy or hypersensitivity to iodine or chlorhexidine
* Active ocular infection
* Contraindication to surgery
* Pregnant women
* Patients residing in nursing homes or prison
* Patients who used antibiotic, antiviral or antifungal eye drops in the week preceding the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Conjunctival composition | 3 days. Conjunctival swabs were taken at baseline and after 3 days of treatment.
  Molecular based method: 16S rRNA gene was sequenced to evaluate ocular microbiota

SECONDARY OUTCOMES:
Patient pain score | Day 3: after 3 days of treatment
  Numerical rating scale, from 0 to 10
Compliance of the patients | Day 3: after 3 days of treatment
  Questionnaire about patients' compliance

CONTACTS AND LOCATIONS:
Overall Officials: Vito Romano, MD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: After completion of the study
Access Criteria: Upon approval of individual sharing request